CLINICAL TRIAL: NCT03845907
Title: Clinical Evaluation of Opto-Acoustic Image Quality With the Gen1B Duplex Probe in Breast Applications
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Data on initial patients sufficient
Sponsor: Seno Medical Instruments Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: GEN1B-01
Record Dates: First submitted 2018-11-07; First posted 2019-02-19 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Unblinded feasibility study in healthy subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Imagio Gen 1B (Active Comparator): Gen 1B duplex probe ultrasound / optoacoustic imaging of the breast and axillary lymph node, with the IMAGIO System and the Gen1B duplex probe
  Interventions: Device: Gen 1B; Device: Gen 1
- Imagio Gen 1 (Active Comparator): Gen 1 duplex probe ultrasound / optoacoustic imaging of the breast and axillary lymph node, with the IMAGIO System
  Interventions: Device: Gen 1B; Device: Gen 1

INTERVENTIONS:
Device: Gen 1B — Diagnostic Ultrasound and Optoacoustic Imaging
Device: Gen 1 — Diagnostic Ultrasound and Optoacoustic Imaging

SUMMARY:
Comparative Evaluation of Gen1B (OA-16-1S) duplex OA/US probe versus Gen1 (OA-16-1) duplex OA/US probe in Healthy Subjects

DETAILED DESCRIPTION:
This study performs the first clinical evaluation of the Gen1B (OA-16-1S) duplex OA/US probe. This probe includes design changes to improve reliability and performance compared to the Gen1 (OA-16-1) duplex OA/US probe. The performance of the Gen1 duplex probe is functionally equivalent to the PIONEER duplex probe (OA-15-3), which was used in previous clinical studies for suspicious breast masses.

ELIGIBILITY:
Inclusion Criteria:

* Has a signed and dated informed consent, prior to initiation of any study-related activities.
* Is at least 18 years of age.
* Is willing to undergo an Imagio imaging evaluation and standard Ultrasound Evaluation of the breast and axillary lymph nodes.
* Is willing and able to comply with protocol-required scans.

Exclusion Criteria:

* Is pregnant or lactating.
* Has a condition or impediment (i.e. insect bites, poison ivy, rash, open wounds, chafing of the skin, scar, tattoos, moles, breast implants within the previous 12 months, etc.) where the duplex probe will come in contact with the subject, which could interfere with the intended field of view.
* Is experiencing photo-toxicity associated with currently taking, or having taken, photosensitizing agents within the previous 72 hours such as sulfa, ampicillin, tetracycline.
* Is currently undergoing phototherapy.
* Has a history of any photosensitive disease (e.g., porphyria, lupus erythematosus) or undergoing treatment for a photosensitive disease and is experiencing photosensitivity.
* Has had an adverse reaction in the past to medical laser procedures, such as laser hair removal or laser tattoo removal.
* Has had a history of contact dermatitis induced by gold or chrome metal contact with skin.
* Has an acute or chronic hematoma and/or acute ecchymosis of the breast.
* Has had prior benign excisional breast biopsy within the past 18 months.
* Has nipple rings that cannot be removed or are not removed during Imagio evaluation.
* Currently has mastitis.
* Has focal pain in the breast.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Treatment-related Events | At end of study, average of six months
  Safety of the Gen 1B duplex Optoacoustic (OA)/ Ultrasound (US) probe in breast applications as compared to Gen 1 with respect to treatment-related events
Diagnostic Image Quality of Gen 1B | At end of study, average of six months
  Independent reader comparison using questionnaire and measurements on artifacts and features of Gen 1 Gen1B probe images for pair wise comparison

SECONDARY OUTCOMES:
Probe performance data comparison across skin types | At end of study, average of six months
  The effect of skin pigmentation using the Fitzpatrick Scale (skin typing test), from Type I (always burns, never tans (palest; freckles) to Type VI never burns (deeply pigmented dark brown to darkest brown) will be used to determine similarities and differences between probes.
Image Quality between probes at reduced laser level | At end of study, average of six months
  OA images with reduced laser level energy will be collected to determine via a 7 point image quality scale, where 1 is poor and 7 is best, which probe produces better images by independent readers

CONTACTS AND LOCATIONS:
Overall Officials: A. Thomas Stavros, MD, Study Director — Seno Medical
Locations (1):
- Seno Medical, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No